CLINICAL TRIAL: NCT02321995
Title: A Quantitative Optical Sensor to Monitor Vascular Physiology; A Healthy Volunteer Study
Status: Completed | Type: Observational
Sponsor: Zenalux Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00057177
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the Zenalux IM1, an optical spectroscopy device with a pressure sensor. The pressure sensor is intended to overcome the inconsistencies attributable to variations in use of the device. This study will involve using the device on healthy volunteers. Three tissue parameters will be used to analyze the pressure effects in two ways: within- and across-subject variability. Measurements will be taken under the tongue and on the inside of the cheek. The device is noninvasive and is approved for preclinical use.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY:

1. There exist significant systematic and random errors in the in vivo spectroscopic measurement of tissue hemoglobin concentrations, blood oxygenation, and scattering coefficient due to uncontrolled probe-to-tissue interface and the lack of a real-time calibration.
2. It is possible to design and engineer a fiber optic sensor to perform accurate and reproducible diffuse reflectance spectroscopy (DRS) for noninvasive quantification of tissue physiology and morphology in vivo. Features such as probe pressure control and instrument self-calibration will improve signal-to-noise ratios by removing user bias from optical measurements.

STUDY OBJECTIVES

1) Evaluation of the pressure sensor in healthy volunteers to determine the minimum contact pressure required for spectroscopic measurements

DESIGN AND PROCEDURES:

Evaluation of the pressure sensor in a volunteer study (n=10)

Informed consent will be obtained from all volunteers. In order to assess the pressure sensor, all research procedures will be repeated twice (once with the aid of the stepper motor and once without the aid of the stepper motor.) For the first five subjects, measurements will be made with the stepper motor first followed by measurements without the stepper motor. The remaining five-subjects will receive the measurements in the reverse order (no stepper motor following by stepper motor). Before the optical measurements, all subjects will be asked to rinse their mouth with a 0.9% saline solution in order to minimize the influence of consumed food. The instrument is high-level disinfected prior to each use in cidex or sterilized by ethylene oxide per standard clinical procedure. Furthermore, it is not anticipated that this device will pose a significant risk to vulnerable populations. The probe will be covered with an optically clear protective sterile sheath and placed in contact with the soft tissue. Reflectance measurements will be taken from each volunteer at up to 5 pressure levels (25, 50, 75, 100, 150 mmHg). At each pressure level 10 spectra will be acquired sequentially. The first measurement will start immediately after the desired probe pressure is reached. This will generate a total of 100 sample and calibration spectra pairs from each subject. This will be repeated on other sites including the tongue, cheek and gums. The sample spectrum will be calibrated using the calibration spectrum collected concurrently. Three tissue parameters will be used to analyze the pressure effects which is described here with [THb] as an example: First, the mean [THb] and its standard deviation will be calculated from the 10 repeat measurements at each pressure for each subject for measurements with and without the stepper motor and plotted against the probe pressure (refer to as THb-P curve). Second, at each pressure level, the [THb] will be plotted against time for each subject and the curve will indicate the temporal response of the tissue under that probe pressure. A series of paired t-tests will be used to identify the contact pressure at which minimal [THb] variance occurs over time (when stepper motor is used). Next, the variance at that contact pressure will be compared to the case without the stepper motor to demonstrate a significant reduction in pressure variance.

The investigators do not anticipate any risks to participants, however, there are a few potential minimal risks such as loss of confidentiality; slight risk of infection; discomfort at the pressure sites; and jaw discomfort as a result of the mouth being opened for several minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer with no presentation of disease (such as no complaints or self-reported oral symptoms or lesions; no cold or flu like symptoms) that would affect the reflective measurements in the oral cavity
* Age 18 or older
* Subjects of all ethnic and gender groups will be included
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects considered in "vulnerable" populations such as children under the age of 18
* Complaint of oral symptoms or lesions
* Current cold or flu like symptoms (self-reported)
* Pregnancy (self-reported by menstrual history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
minimum contact pressure required for spectroscopic measurements | at the time the optical measurements are collected

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dewhirst, DVM, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States